CLINICAL TRIAL: NCT05002465
Title: Clinical Use of 68Ga Prostate Specific Membrane Antigen-11 Positron Emission Tomography With Computed Tomography in Diagnosing, Staging and Restaging Prostate Cancer
Brief Title: Clinical Use of 68Ga PSMA-11 PET/CT in Diagnosing, Staging and Restaging Prostate Cancer
Status: No longer available | Type: Expanded Access
Sponsor: Dana Mathews (Other)
Responsible Party: Sponsor-Investigator, Dana Mathews, Professor, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Other Study IDs: STU-2021-0291
Record Dates: First submitted 2021-07-27; First posted 2021-08-12 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer; Prostate Cancer Metastatic; Prostate Cancer Recurrent
Keywords: Gallium-68; PSMA-11; PET/CT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: 68Ga-PSMA-11 — Injection of 68Ga PSMA-11
Procedure: Positron Emission Tomography/Computed Tomography — PET/CT scan after 68Ga PSMA-11 injection
  Other Names: PET/CT

SUMMARY:
The purpose of this protocol is to provide 68Ga Prostate Specific Membrane Antigen-11 (68Ga PSMA-11) for clinical use in the diagnosis, staging and restaging of prostate cancer using Positron Emission Tomography with Computed Tomography (PET/CT) prior to its full local Federal Drug Administration (FDA) approval. Extensive research has shown that 68Ga PSMA-11 PET/CT offers higher detection rate of metastatic disease in prostate cancer than the current standard of care usually used in staging and restaging prostate cancer.

DETAILED DESCRIPTION:
68Ga PSMA-11 PET/CT offers higher detection rate of metastatic disease in prostate cancer than the current standard of care of computed tomography (CT), magnetic resonance imaging (MRI), and bone scintigraphy usually used in staging and restaging prostate cancer. Furthermore, 68Ga PSMA-11 PET/CT offers a higher detection rate of primary and metastatic prostate cancer compared to other available radiotracers used for prostate cancer. It additionally offers enhanced imaging characteristics of greater sensitivity at lower prostate specific antigen (PSA) values and higher target to background ratios than currently available radiotracers. For these reasons, we feel that expanded access to 68Ga PSMA-11 offers better patient care at comparable cost to standard imaging.

The population to be treated consists of men in whom metastatic or recurrent prostate cancer is suspected. Patients will be recruited primarily from the clinical practices of the University of Texas Southwestern Medical Center (UTSW) and Parkland Health and Hospital System. Additional patients may be referred for recruitment from physicians outside UTSW.

Each patient will receive an IV injection of 68Ga PSMA-11 as a bolus intravenous injection. Depending on patient medical history and Radiology physician preference, the patient may also be injected with 20 milligrams (mg) of furosemide to encourage urination, and the patient will void immediately prior to getting on the scan table. Patients will be scanned on a PET/CT scanner. The patient will be positioned with arms elevated above the head.

ELIGIBILITY:
Inclusion Criteria:

* One of the following:

  1. Patients with suspected recurrence based on elevated serum prostate specific antigen (PSA) level.
  2. Patients with suspected metastasis who are candidates for initial definitive therapy.
  3. Patients with metastatic prostate cancer, for whom Lutetium-177 vipivotide tetraxetan PSMA-directed therapy is indicated.
* Patients must be able to lie still for approximately 20 - 40 minutes for the PET/CT scans.
* Patients must be deemed medically stable by their treating physician.
* Patients must have the ability and willingness to sign a written informed consent.

Exclusion Criteria:

* Patients must not weigh more than the maximum weight limit for the PET/CT scanner table (> 225 kilograms or 500 pounds).
* Patients must not have history of allergic reactions attributed to compounds of similar chemical or biologic composition to 68Ga PSMA-11.
* Patients must not be claustrophobic.

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes

CONTACTS AND LOCATIONS:
Overall Officials: Orhan K Oz, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States